CLINICAL TRIAL: NCT07320872
Title: Correlation Between Vaspin Gene Polymorphism and Serum Vaspin Levels in Psoriasis Vulgaris and Its Relation to Pathogenesis and Risk of the Disease
Brief Title: Correlation Between Vaspin Gene Polymorphism and Serum Vaspin Levels in Psoriasis Vulgaris
Status: Recruiting | Type: Observational
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Ola Mahmoud Elqousy, Specialist at Dermatology, Venereology and Andrology Department, Aswan University
Other Study IDs: Psoriasis Vulgaris Vaspin Gene
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-08

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sampling withdrawn from both healthy and control groups subjected for DNA extraction and SNP genotyping of vaspin gene polymorphism by real time - PCR. and Serum samples will be also taken to detect the serum level of vaspin concentrations by ELISA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Psoriasis Patients: About 30 patients suffering from Psoriasis Vulgaris will subject to vaspin gene polymorphism measure and Assessment of the disease severity will be performed by using Psoriasis area and severity index score (PASI score) for all patients.
  Interventions: Biological: vaspin gene polymorphism
- Group B: Control Group: About 30 healthy participants will share as A control Group
  Interventions: Biological: vaspin gene polymorphism

INTERVENTIONS:
Biological: vaspin gene polymorphism — to detect the correlation between vaspin gene polymorphism and serum vaspin levels among psoriasis patients.
  * To detect the relationship between the risk of psoriasis and the vaspin gene polymorphism.
  * To detect correlation between vaspin gene polymorphism and the severity of psoriasis.
  Other Names: Serum Vaspin Levels

SUMMARY:
Psoriasis is a common immune-mediated inflammatory skin disease affecting at least 100 million individuals worldwide. In Egypt, the prevalence of psoriasis ranges between 0.19% and 3% of the Egyptian people.

It is associated with poor quality of life, reduced life expectancy and multimorbidity including psoriatic arthritis, obesity and cardiovascular disease.

Vaspin (VASP, SERPIN 12) is a recently discovered adipokine that has been isolated from the visceral adipose tissue of a rat model of type 2 diabetes. It is coded by the gene SERPNA12 located on the long arm of chromosome 14q32.13 and consists of six exons and five introns.

DETAILED DESCRIPTION:
Psoriasis can present at any age. However, the disease onset appears to follow a bimodal distribution, peaking around 20-30 years of age and again around 50-60 years of age.

Psoriasis is a common skin disease characterized clinically by formation of erythematous and scaly plaques at different sites affecting mainly the extensor prominences, scalp, the lumbosacral area and the sites of trauma. It is a lifelong disease with spontaneous remissions and exacerbations.

The exact etiology is unknown, but it is considered to be an autoimmune disease mediated by T lymphocytes. It is considered the most prevalent T-cell-mediated inflammatory disease in human beings, in which, keratinocytes in focal skin regions are stimulated to proliferate with activation of the immune system mediated by primed T-lymphocytes.

There is an association of HLA antigens seen in many psoriatic patients, particularly in various racial and ethnic groups. Familial occurrence suggests its genetic predisposition .

The pathophysiology of psoriasis involves infiltration of the skin by activated T cells which stimulate the proliferation of keratinocytes. This dysregulation in keratinocyte turnover results in the formation of thick plaques. Other associated features include epidermal hyperplasia and parakeratosis. There are several treatment options available for mild psoriasis, including topical corticosteroids, vitamin D analogs, calcineurin inhibitors, keratolytics, and targeted phototherapy.

More severe disease might require systemic therapy, including phototherapy, acitretin, methotrexate, cyclosporine, or biologic therapy. Psoriasis is accompanied by comorbidities such as obesity, diabetes, and metaboloic syndrome. Although the pathogenesis is still unknown, systemic inflammation caused by adipokines released from visceral adipose tissue is thought to play a role .

Adipokines are various bioactive polypeptides produced and released by adipose tissue. Adipokines are thought to play an important role in the pathogenesis of obesity-related diseases such as insulin resistance, hypertension, inflammation, and metabolic disorders.

Vaspin (visceral adipose tissue-derived serine protease inhibitor also called Serpin A12), It belongs to the serpin group of proteins and is a serine protease inhibitor produced from visceral adipose tissue.Vaspin consists of 415 amino acids and weighing 47-kDa .

Vaspin is an adipokine with recently described anti-inflammatory properties. It has been reported to be expressed in various tissues, such as skin, liver, stomach and pancreas, in addition to adipose tissue in humans . The main source of vaspin in human skin was found to be keratinocytes. Vaspin in the skin is associated with the differentiation of keratinocytes and suppresses the expression of inflammatory mediators.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed cases or stopped treatment of at least 6 months of psoriasis patients.
* Pateints with any age and gender.

Exclusion Criteria:

* Pregnancy and lactation.
* Patients with chronic diseases: cardiac diseases, hepatic disorders, chronic renal failure or malignancies.
* Patients with associated inflammatory disease such as infections and autoimmune diseases.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include (30) psoriasis patients and (30) normal control. and will be conducted on psoriasis patients and the healthy persons whom will be selected from the outpatient clinic of the Dermatology, Venereology, and Andrology Department, at Aswan University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08-10 (Actual); Primary Completion 2026-08-10 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Detection of vaspin gene polymorphism | 12 Months
  Assessment of vaspin gene polymorphism in psoriasis patients to determine the disease severity

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa Adam Ali El Taieb, Professor, Study Chair — Dermatology, Venereology and Andrology.Faculty of Medicine, Aswan University; Hoda Soltan Sherkawy El Bakry, Lecturer, Study Director — Medical biochemistry,Faculty of Medicine,Aswan University
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided